CLINICAL TRIAL: NCT06952010
Title: A Phase 1 Study of XB628 in Participants With Recurrent Advanced or Metastatic Solid Tumors
Brief Title: A Study of XB628 in Participants With Recurrent Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XB628-101
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Advanced Solid Tumor; Metastatic Solid Tumor; Immune Sensitive Tumor
Keywords: XB628; Solid tumor; Advanced solid tumor; Metastatic solid tumor; Immune sensitive tumor; PD-L1
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- XB628 (Experimental): Group(s) of participants with recurrent advanced or metastatic solid tumors will receive escalating dose levels doses of XB628.
  Interventions: Biological: XB628

INTERVENTIONS:
Biological: XB628 — Intravenous infusion(s)

SUMMARY:
This is a phase 1, first-in-human, open-label, dose-escalation study of XB628, a first-in-class bispecific antibody natural killer (NK) cell engager that targets NK group 2 member A (NKG2A), an inhibitory receptor on NK cells, and programmed cell death-ligand 1 (PD-L1).

DETAILED DESCRIPTION:
This study consists of a Dose-Escalation Stage. The Dose-Escalation Stage is designed to determine the maximum tolerated dose (MTD) and/or recommended dosage(s) for expansion (RDE[s]) of XB628 as a single agent.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Minimum life expectancy of ≥ 12 weeks.
* Have a recurrent advanced or metastatic solid tumor that is histologically or cytologically confirmed.
* Adequate organ and marrow function.
* Not amenable to curative treatment with surgery or radiation.
* Received at least 1 line of prior systemic anticancer therapy in the recurrent or metastatic setting.
* Acceptable alternative therapy was received, refused, intolerable, or no longer effective.
* Capable of understanding and complying with the protocol requirements and provide signed informed consent according to the protocol and local requirements.

Exclusion Criteria

* Primary brain tumors or known active brain metastases.
* Major surgery (eg, gastrointestinal surgery, removal or biopsy of brain metastasis) within 4 weeks before the first dose of study treatment.
* Received radiation therapy within 1 week before the first dose of study treatment or clinically relevant ongoing complications from prior radiation therapy.
* Received prior therapy targeting NK cells (eg, monalizumab).
* A woman of childbearing potential has a positive serum pregnancy test within 7 days prior to study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLTs) | 21 days
Number of Participants with Serious Adverse Events (SAEs), Treatment-emergent Adverse Events (TEAEs), and Adverse Events (AEs) Leading to Dose Withholding, Treatment Discontinuation, or Death | 27 months

SECONDARY OUTCOMES:
Area Under the Concentration-time Curve (AUC) of XB628 | 25 months
Maximum Plasma Concentration (Cmax) of XB628 | 25 months
Time to Maximum Concentration (Tmax) of XB628 | 25 months
Elimination Half-life (T1/2) of XB628 | 25 months
Apparent Clearance (CL/F) of XB628 | 25 months
Trough Concentration (Ctrough) of XB628 | 25 months
Number of Participants with Antidrug Antibody (ADA) Response to XB628 | 25 months
Objective Response Rate (ORR) | 27 months
Duration of Response (DOR) | 27 months
RDE for XB628 | 25 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Exelixis
Locations (10):
- United States (10):
  - Exelixis Site #5, San Francisco, California
  - Exelixis Site #4, New Haven, Connecticut
  - Exelixis Clinical Site #8, Tampa, Florida
  - Exelixis Clinical Site #10, Boston, Massachusetts
  - Exelixis Site #6, St Louis, Missouri
  - Exelixis Site #7, New York, New York
  - Exelixis Clinical Site #1, Hickory, North Carolina
  - Exelixis Clinical Site #3, Nashville, Tennessee
  - Exelixis Clinical Site #9, Houston, Texas
  - Exelixis Clinical Site #2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No